CLINICAL TRIAL: NCT02350803
Title: Dose Use of Rigid Fixation After Removing the Distraction Device Reduce the Anterior-posterior Relapse or Not?
Brief Title: Does Use of Rigid Fixation After Removing Distraction Osteogenesis Device Reduce the Relapse?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Reza Tabrizi, Assistant professor of oral and maxillofacial surgery, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUDO-1394
Record Dates: First submitted 2015-01-16; First posted 2015-01-30 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Cleft Palate; Maxillary Hypoplasia; Maxillary Retrognathism
Keywords: distraction osteogenesis; mini plate; Lefort 1 osteotomy
MeSH Terms: conditions — Cleft Palate; Retrognathia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- distraction osteogenesis (Placebo Comparator): treatment of maxillary deficiency was done just by distraction osteogenesis and no mini plate was used after removal of distractor
- distraction osteogenesis+ mini plate (Active Comparator): treatment of maxillary deficiency was done just by distraction osteogenesis and after removal of distractor 4 mini plate L shaped was used after removal of distractor as an intervention
  Interventions: Device: mini plate

INTERVENTIONS:
Device: mini plate — in the intervention group, 4 L shaped titanium mini plates with 16 screws were fixed immediately after distraction phase and removal of distraction ossteogenesis to prevent the relapse after distraction
  Arms: distraction osteogenesis+ mini plate

SUMMARY:
patients were enrolled by the inclusion criteria and were undergo lefort 1 maxillary osteotomy. after the latency phase the distraction was done in anterior- posterior vector. patients were divided by randomized allocation in 2 groups. in group 1 the distractor was removed after consolation phase, and in group 2 fixation devices were placed immediately after removal of distractors. data regarding relapse were analyzed by lateral cephalogram X-ray taken in 3 different phases of the trial. change of occlusal plane and the "A point" of the cephalometric analysis were determined as reference point of the study.

DETAILED DESCRIPTION:
All patients were undergo maxillary Lefort 1 osteotomy with intra oral distractors bilaterally. The latency phase was considered 5 days for all of them. Distraction was done in the anterior- posterior vector with 1 mm/day rate. In group 1 distraction devices were removed after finishing distraction and a 3 months consolation, in group 2 fixation devices (4 L shaped miniplates with 16 screws) were placed immediately after removing distractors.

The amount of horizontal and vertical relapse were determined in the "A point" 2 years after finishing distraction.

By using lateral cephalogram X-ray as a raw data base, taken in 3 occasions: preoperatively, immediately after finishing consolation phase and removing distractor with placing fixation devices or without them and 2 years postoperatively in every subject. Relevant skeletal points were determined and digitized to evaluate 2-dimensional skeletal changes during and after surgery and to subsequently determine the amount of relapse. The same X-ray machine and settings were used for all cephalograms.Patients were stabilized in the lateral Cephalogram unit (Planmeca, ProMax, Helsinki-Finland) using Cephalostat. With the position of the patients with their head oriented at 90 degree angle to the X-Ray beam at a distance of 5ft from the tube. The jaws were in maximum intercuspation, tip of the tongue behind the upper incisor teeth and lips in relaxed position. The receptor (CR, Konica Minolta medical imaging, USA) was placed 15 inches from the head. This is a standard under which all cephalometric radiographs are taken. It ensures that radiographs, taken in different times, are directly comparable.

Radiographic exposures were 60-80 Kvp, 10-15 mA, and 16-32 sec, and repeated for each case in three occasions.

The radiographs were processed in laser readout processor special for mentioned CR system. PACS. A DICOM system used for saving and transferring the images.

All Lateral cephalograms were traced by hand and digitized, superimposed and evaluated by the same examiner. The tracings were rechecked by another examiner.

ELIGIBILITY:
Inclusion Criteria:

patients need lefort 1 maxillary advancement more than 8 mm and have presurgical orthodontic preparation

Exclusion Criteria:

patients with cleft lip and alveolar cleft ,traumatic patients ,patients with previous orthognathic surgery in the maxilla and edentulous patients

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2013-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
"A point" of lateral cephalometry X-ray | 2 years after finishing the distraction
  "A point" is used to determine the horizontal and vertical relapse

SECONDARY OUTCOMES:
occlusal plane | 2 years after distraction is finished
  changes in occlusal plane is determine to assess the amount of relapse

CONTACTS AND LOCATIONS:
Overall Officials: Reza Tabrizi, DMD, Study Director — Shiraz University of Medical Sciences; Touba Karagah, DMD, Principal Investigator — Shiraz University of Medical Sciences; Negin Matini, DMD, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- shiraz University of medical sciences, Shiraz, Fars, Iran